CLINICAL TRIAL: NCT02085889
Title: Fructose and Lactose Intolerance and Malabsorption: the Relationship Between Metabolism and Symptoms in Functional Gastrointestinal Disorders
Brief Title: Fructose and Lactose Intolerance and Malabsorption in Functional Gastrointestinal Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brain-Gut Research Group (Other)
Responsible Party: Principal Investigator, Clive H Wilder-Smith, MD, Principle Investigator, Brain-Gut Research Group
Other Study IDs: BGRG-2415b
Record Dates: First submitted 2014-03-10; First posted 2014-03-13 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Functional Gastrointestinal Disorders; Lactose Intolerance; Fructose Intolerance
MeSH Terms: conditions — Gastrointestinal Diseases; Lactose Intolerance; Fructose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, urine and stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- food intolerance: lactose intolerance fructose intolerance neither intolerance
  Interventions: Other: no intervention: observational study

INTERVENTIONS:
Other: no intervention: observational study — observational

SUMMARY:
Background: The association of fructose and lactose intolerance and malabsorption with the symptoms of different functional gastrointestinal disorders (FGID) is unclear. The mechanisms behind the multi-organ symptoms remain unclear. Both FGID and saccharide intolerances are common (>10% of any given population). Dietary modification based on intolerance diagnostics could provide an effective treatment for FGID, which are otherwise difficult to treat.

Aim: To investigate the prevalence and interrelationships of fructose and lactose intolerance (symptom induction) and malabsorption (breath test gas production) and their association with clinical GI as well as non-GI symptoms in FGID and the outcome of standard dietary intervention. Mechanisms related to symptom genesis will be investigated using metabolomic analysis of plasma and urine by gas chromatography/time-of-flight mass spectrometry (GC/TOFMS).

Methods: Fructose and lactose intolerance (defined by positive symptom index) and malabsorption (defined by increased hydrogen/methane) will be determined in successive male and female FGID patients in a single center using breath-testing. Symptoms will be recorded using standardised questionnaires and the Rome III criteria. The prevalence of the intolerances in the different FGID subgroups and the associations between breath testing results, clinical symptoms and the outcome of dietary modification will be assessed. Factors predictive of the outcome of dietary modulation will be screened for. GC/TOFMS will be used to assess the human and microbial metabolome in urine and plasma.

ELIGIBILITY:
Inclusion criteria:

* Patients with functional GI disorders according to ROME 3 criteria
* Without evidence of organic disease by standardised testing in GI practice.

Exclusion criteria:

* Current or relevant history of organic disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Successive patients referred to our gastroenterology practice with functional GI disorders according to ROME 3 criteria.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number with adequate symptom relief | 6-12 weeks
  adequate symptom relief in response to reduction of fermentable sugars

SECONDARY OUTCOMES:
Association between adequate symptom relief and test variables | 6-12 weeks
  association between demographic, breath test and metabolomic factors and adequate relief due to dietary modification

CONTACTS AND LOCATIONS:
Overall Officials: Clive Wilder-Smith, MD, Principal Investigator — Brain-Gut Research Group
Locations (1):
- Gastoenterology Group Practice, Bern, Switzerland

REFERENCES:
- [Derived] Wilder-Smith CH, Drewes AM, Materna A, Olesen SS. Extragastrointestinal Symptoms and Sensory Responses During Breath Tests Distinguish Patients With Functional Gastrointestinal Disorders. Clin Transl Gastroenterol. 2020 Aug;11(8):e00192. doi: 10.14309/ctg.0000000000000192. PMID 32955198
- [Derived] Wilder-Smith CH, Olesen SS, Materna A, Drewes AM. Fermentable Sugar Ingestion, Gas Production, and Gastrointestinal and Central Nervous System Symptoms in Patients With Functional Disorders. Gastroenterology. 2018 Oct;155(4):1034-1044.e6. doi: 10.1053/j.gastro.2018.07.013. Epub 2018 Sep 3. PMID 30009815
- [Derived] Wilder-Smith CH, Olesen SS, Materna A, Drewes AM. Breath methane concentrations and markers of obesity in patients with functional gastrointestinal disorders. United European Gastroenterol J. 2018 May;6(4):595-603. doi: 10.1177/2050640617744457. Epub 2017 Nov 15. PMID 29881615